CLINICAL TRIAL: NCT01034813
Title: Assessment of Joint Range of Motion and Cutaneous Functional Unit Recruitment: Association With Burn Scar Characteristics
Brief Title: Joint Range of Motion in Burn Scars
Status: Terminated | Type: Observational
Why Stopped: New PI discovered that some of previously collected data may not be accurate
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: H-09-039
Record Dates: First submitted 2009-12-16; First posted 2009-12-18 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Contractures Resulting From Burn Scar Tissue
Keywords: contractures, range of motion, scar formation
MeSH Terms: conditions — Contracture

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Burn Range of motion: burn patients with hypertropic scar
- control range of motion: control subjects without scaring

SUMMARY:
The purpose of this study is to determine the relationship between cutaneous functional unit(CFU)recruitment throughout the available active range of motion of a prescribed joint in normal subjects and patients with burn scars. Specifically, this study will determine if differences in CFU recruitment exist between normal subjects and individuals with burn scars at the dorsal hand, dorsal or volar forearm, or anterior or posterior arm during active range of motion of the MCP joint during flexion, or the wrist or elbow during flexion or extension, respectively.

DETAILED DESCRIPTION:
Specific Aim #1: To establish the relationship between joint position and skin recruitment, expressed as the percentage of CFU recruited during active ROM, in patients with burn scars and normal controls.

Specific Aim #2: To establish the within-day and between-day reliability of percent CFU estimation and absolute skin recruitment, measured in millimeters from a fixed reference, during active ROM for a specified joint.

Specific Aim #3: To establish the relationship between scar height, measured by diagnostic ultrasound, scar cross-sectional area, and percent CFU recruitment in individuals with burn scar.

Specific Aim #4: To determine whether the amount of skin recruitment, expressed as the percent of the CFU recruited during active ROM, is differentially affected by burn scar.

Ho: There is no difference in the percent CFU recruited at the completion of active range of motion at a specified joint between individuals with burn scars and normal controls.

Ha: Individuals with burn scars recruit a greater percentage of the CFU in order to obtain maximal range of motion at a specified joint.

Specific Aim #5: To determine whether the timing of skin recruitment, expressed as the initiation of skin movement within a CFU relative to joint position during active ROM, is differentially affected by burn scar.

Ho: There is no difference in the initiation of skin movement within a CFU relative to joint position during active ROM at a specified joint between individuals with burn scars and normal controls.

Ha: In individuals with burn scars in a given CFU, skin movement farther from the joint axis occurs earlier in the range of motion compared to controls.

Specific Aim #6: To determine whether skin extensibility within a CFU during active ROM of a specified joint is differentially affected by burn scar.

Ho: There is no difference skin extensibility within a CFU during active ROM of a specified joint between individuals with burn scars and normal controls.

Ha: In individuals with burn scars in a given CFU, skin near the joint axis undergoes greater deformation (stretch) as range of motion at the joint increases compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria include: 1) male or female burn survivors between the ages of 18 and 60, 2) an area of scar covering at least fifty percent of the CFU of interest, 3) control subjects must have full active range of motion of the metacarpal phalangeal joints, wrist and elbow according to published normative references and be free of any history neuromusculoskeletal injury within the last three years that involved the joints of interest.

Exclusion Criteria:

* Exclusion Criteria include: 1)burn survivors with an area of scar of less than fifty percent of the CFU of interest, 2) burn survivors with a history of orthopedic trauma to the upper extremity (i.e. sprain within the last 24 months, history of fracture, or history of joint dislocation), 3) control subjects with a history of upper extremity trauma or injury, 4) control subjects with the presence of scar tissue covering an area of more than one percent of the CFU of interest, 5) any potential subject with a history or rheumatoid arthritis, osteoarthritis affecting the extremity of interest, peripheral nerve injury of the extremity of interest, or systemic disorder affecting joint range of motion of the upper extremity.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Military and civilian burn patients.Control population will be individuals without upper extremity injury.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2010-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Range of motion | 3-5 days

SECONDARY OUTCOMES:
Scar Hypertrophy | 3--5 days

CONTACTS AND LOCATIONS:
Overall Officials: William S Dewey, PT, CHT, Principal Investigator — United States Army Institute of Surgical Research
Locations (1):
- USAISR, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Nedelec B, Correa JA, Rachelska G, Armour A, LaSalle L. Quantitative measurement of hypertrophic scar: interrater reliability and concurrent validity. J Burn Care Res. 2008 May-Jun;29(3):501-11. doi: 10.1097/BCR.0b013e3181710881. PMID 18388576